CLINICAL TRIAL: NCT01227135
Title: CHOICES: A Randomized Phase II Trial of Imatinib (IM) Versus Hydroxychloroquine (HCQ) and IM for Patients With Chronic Myeloid Leukemia (CML) in Major Cytogenetic Response (MCyR) With Residual Disease Detectable by Quantitative Polymerase Chain Reaction (Q-PCR).
Brief Title: Imatinib Mesylate With or Without Hydroxychloroquine in Treating Patients With Chronic Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lynn McMahon (Other)
Collaborators: Medical Research Council (Other Government); CRUK Trials unit Glasgow (Unknown)
Responsible Party: Sponsor-Investigator, Lynn McMahon, Project Manager, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000686729; CRUK-H135; ISRCTN-61568166; EUDRACT-2009-014373-41; EU-21078
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Hydroxychloroquine; Imatinib Mesylate; Cytogenetic Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: hydroxychloroquine
Drug: imatinib mesylate
Genetic: cytogenetic analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as hydroxychloroquine, may stimulate the immune system in different ways and stop cancer cells from growing. It is not yet known whether imatinib mesylate is more effective when given with or without hydroxychloroquine in treating patients with chronic myeloid leukemia.

PURPOSE: This randomized phase II trial is studying the side effects of giving imatinib mesylate with or without hydroxychloroquine and to see how well it works in treating patients with chronic myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if imatinib mesylate versus hydroxychloroquine (HCQ) and imatinib mesylate is more effective in terms of BCR/ABL levels in patients with chronic myeloid leukemia in major cytogenetic response (MCyR) with residual BCR/ABL-positive cells detectable by quantitative polymerase chain reaction after at least one year of imatinib mesylate treatment.
* To determine the safety and tolerability of this regimen in these patients.

Secondary

* To determine whether the introduction of HCQ influences imatinib mesylate plasma levels.
* To determine if whole blood HCQ levels achieved in combination with imatinib mesylate are in the expected range.
* To determine if HCQ inhibits autophagy in vivo.
* To evaluate the effects of this regimen on residual BCR/ABL-positive primitive progenitors.

OUTLINE: This is a multicenter study. Patients are stratified according to baseline polymerase chain reaction (PCR) level (< 3 logs below baseline vs ≥ 3 logs below baseline), time on imatinib mesylate (12 to < 24 months vs 24 to < 36 months), imatinib mesylate dose (< 400 mg vs 400 mg to < 600 mg vs 600 mg to 800 mg), and center. Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive oral imatinib mesylate daily. Treatment repeats every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.
* Arm B: Patients receive oral imatinib mesylate daily and oral hydroxychloroquine (HCQ) twice daily. Treatment repeats every 4 weeks for up to 12 months in the absence of disease progression or unacceptable toxicity.

In both arms, patients may then receive oral imatinib mesylate daily for another 12 months during the follow up period of this study.

Consenting patients undergo blood sample and bone marrow collection at baseline, during, and after completion of study therapy for pharmacologic and other laboratory studies.

After completion of study treatment, patients are followed up at 3, 6, 9, and 12 months.

Peer Reviewed, Funded by MRC and supported by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic myeloid leukemia (CML) in chronic phase (CP)
* Has been treated with imatinib mesylate for at least 1 year

  * Receiving a stable dose for ≥ 6 months prior to randomization
* Achieved at least major cytogenetic response (MCyR) and continues to be BCR/ABL-positive by quantitative polymerase chain reaction (Q-PCR)
* Must have a fusion gene present that can be monitored by Q-PCR

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³ (stable and within normal range for ≥ 2 months)
* Platelet count ≥ 100,000/mm³ (stable and within normal range for ≥ 2 months)
* Serum albumin > 3 g/dL
* AST and/or ALT ≤ 2.5 times upper limit of normal (ULN)
* Serum bilirubin ≤ 1.5 times ULN
* Serum creatinine ≤ 1.5 times ULN OR 24-hour creatinine clearance ≥ 50 mL/min
* Serum potassium ≥ lower limit of normal with or without replacement therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception (including a barrier method [i.e., condom]) during and for 3 months after completion of study therapy
* No impaired cardiac function, including any of the following:

  * QTc > 450 msec on screening ECG
  * Congenital long QT syndrome
  * History or presence of sustained ventricular tachycardia
  * History of ventricular fibrillation or Torsades de pointes
  * NYHA class III-IV congestive heart failure
  * Uncontrolled hypertension
* No severe gastrointestinal (GI) disorder, uncontrolled epilepsy, known glucose-6-phosphate dehydrogenase (G6PD) deficiency, known porphyria, moderate or severe psoriasis, known myasthenia gravis, or other concurrent severe and/or uncontrolled medical conditions
* No preexisting maculopathy of the eye
* No significant history of noncompliance to medical regimens or the inability to grant a reliable informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy, investigational drug, or major surgery and recovered
* More than 6 months since change in imatinib mesylate dose
* No other concurrent anticancer therapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of treatment "successes" defined as patients who have at least 0.5 log reductions or more in their 12-month PCR level from baseline

SECONDARY OUTCOMES:
Proportion of treatment "successes" at 24 months
Molecular response at 12 and 24 months (complete response, major response, or no response)
Proportion of patients with progression at 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Holyoake, MD, Principal Investigator — Gartnavel General Hospital
Locations (3):
- United Kingdom (3):
  - Royal Liverpool University Hospital, Liverpool, England
  - Imperial College London, London, England
  - Gartnavel General Hospital, Glasgow, Scotland